CLINICAL TRIAL: NCT00652392
Title: A 12 Week, Randomized, Double-Blind, Double-Dummy, Placebo and Active-controlled Study of Symbicort pMDI Administered Once Daily in Adults and Adolescents With Asthma - STEM
Brief Title: Efficacy of Symbicort pMDI Administered Once Daily in Adolescents and Adults During 12 Weeks - STEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-039-0726; D5896C00726
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: asthma; adolescents; adults; Symbicort; budesonide/formoterol; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol
- 2 (Placebo Comparator)
  Interventions: Drug: budesonide and placebo

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: budesonide and placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare a dose of Symbicort taken once daily with other dosage regimens of Symbicort , budesonide and placebo for the treatment of asthma in adolescents and adults

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma and baseline lung function tests as determined by the protocol
* Required and received treatment with inhaled corticosteroids within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Severe asthma
* Has required treatment with any non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in protocol or requires treatment with beta-blockers

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2003-04; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Change in evening PEF | Daily throughout the 12 week treatment period

SECONDARY OUTCOMES:
Lung function, asthma symptoms, use of rescue medication and parent/caregiver/physician reported outcomes | Daily throughout the 12 week treatment period
Health-related quality of life | 4 assessments within 12 week treatment period
Routine safety assessments | 4 assessments within 12 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca

REFERENCES:
- [Derived] Berger WE, Bleecker ER, O'Dowd L, Miller CJ, Mezzanotte W. Efficacy and safety of budesonide/formoterol pressurized metered-dose inhaler: randomized controlled trial comparing once- and twice-daily dosing in patients with asthma. Allergy Asthma Proc. 2010 Jan-Feb;31(1):49-59. doi: 10.2500/aap.2010.31.3309. PMID 20167145